CLINICAL TRIAL: NCT00046345
Title: Atazanavir for HIV Infected Individuals: An Early Access Program
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Other Study IDs: AI424-900
Record Dates: First submitted 2002-09-26; First posted 2002-09-30 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

INTERVENTIONS:
Drug: Atazanavir (BMS-232632)

SUMMARY:
The purpose of this clinical research study is to provide atazanavir to patients infected with human immunodeficiency virus (HIV) whose antiviral medications are no longer working to control HIV activity within the body and who are unable to create a new treatment regimen using other available anti-HIV drugs, because of either side effects or treatment failure previously taken. The safety of this treatment will also be studied.

ELIGIBILITY:
Key inclusion criteria:

* Patients eligible for inclusion into the EAP are those that are a virologic failure due to resistance, intolerance and/or adherence problems with current anti-HIV medications;
* OR have multiple toxicities or intolerance to their anti-HIV medication but are not a virologic failure;
* OR have severe elevated lipids in the blood (e.g., cholesterol, triglycerides) that do not respond to lipid-lowering medication.

Key exclusion Criteria:

* Restrictions apply regarding the use of atazanavir with specific medications which may have a potential to cause possible side effects when taken together.
* Patients will also be excluded for any of the following reasons: 1) pregnancy or breast feeding, 2) elevated liver enzymes, 3) significant cardiovascular disease, or 4) other restrictions as indicated in the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-05; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (163):
- United States (161):
  - Local Institution, Hobson City, Alabama
  - Local Institution, Anchorage, Alaska
  - Local Institution, Phoenix, Arizona
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Bakersfield, California
  - Local Institution, Berkeley, California
  - Local Institution, Beverly Hills, California
  - Local Institution, El Cajon, California
  - Local Institution, Fairfield, California
  - Local Institution, Fontana, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Glendale, California
  - Local Institution, Harbor City, California
  - Local Institution, Lancaster, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Mill Valley, California
  - Local Institution, Newport Beach, California
  - Local Institution, Oakland, California
  - Local Institution, Palm Springs, California
  - Local Institution, Palo Alto, California
  - Local Institution, Panorama City, California
  - Local Institution, Paramount, California
  - Local Institution, Sacramento, California
  - Local Institution, San Bernardino, California
  - Local Institution, San Diego, California
  - Local Institution, San Francisco, California
  - Local Institution, San Jose, California
  - Local Institution, San Mateo, California
  - Local Institution, San Rafael, California
  - Local Institution, Santa Ana, California
  - Local Institution, Santa Rosa, California
  - Local Institution, Sherman Oaks, California
  - Local Institution, Sunnyvale, California
  - Local Institution, Tarzana, California
  - Local Institution, West Hills, California
  - Local Institution, Woodland Hills, California
  - Local Institution, Denver, Colorado
  - Local Institution, Wheat Ridge, Colorado
  - Local Institution, Hartford, Connecticut
  - Local Institution, Meriden, Connecticut
  - Local Institution, Norwalk, Connecticut
  - Local Institution, Rockville, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Bay Pines, Florida
  - Local Institution, Bradenton, Florida
  - Local Institution, Daytona Beach, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Fort Myers, Florida
  - Local Institution, Gainesville, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Key West, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Miami Beach, Florida
  - Local Institution, North Miami Beach, Florida
  - Local Institution, North Palm Beach, Florida
  - Local Institution, Oakland Park, Florida
  - Local Institution, Pensacola, Florida
  - Local Institution, Plantation, Florida
  - Local Institution, Pompano Beach, Florida
  - LOcal Instituton, Sarasota, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Vero Beach, Florida
  - Local Institution, Winter Haven, Florida
  - Local Institution, Winter Park, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Decatur, Georgia
  - Local Institution, Jesup, Georgia
  - Local Institution, Macon, Georgia
  - Local Institution, Tucker, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Kahului, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Joliet, Illinois
  - Local Institution, Springfield, Illinois
  - Local Institution, Evansville, Indiana
  - Local Institution, Munster, Indiana
  - Local Institution, Kansas City, Kansas
  - Local Institution, Topeka, Kansas
  - Local Institution, Paducah, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Portland, Maine
  - Local Institution, Baltimore, Maryland
  - Local Institution, Bethesda, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Hyannis, Massachusetts
  - Local Institution, Provincetown, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Berkley, Michigan
  - Local Institution, Grand Rapids, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Rochester, Minnesota
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Reno, Nevada
  - Local Institution, Camden, New Jersey
  - Local Institution, Elizabeth, New Jersey
  - Local Institution, Englewood, New Jersey
  - Local Institution, Hackensack, New Jersey
  - Local Institution, Hoboken, New Jersey
  - Local Institution, Neptune City, New Jersey
  - Local Institution, Newark, New Jersey
  - Local Institution, Union, New Jersey
  - Local Institution, Voorhees Township, New Jersey
  - Local Institution, West Orange, New Jersey
  - Local Instituton, Westfield, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Santa Fe, New Mexico
  - Local Institution, Brooklyn, New York
  - Local Institution, Elmira, New York
  - Local Institution, Mount Vernon, New York
  - Local Institution, New Hyde Park, New York
  - Local Institution, New York, New York
  - Local Institution, Rochester, New York
  - Local Institution, Southampton, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Valhalla, New York
  - Local Institution, Asheville, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Greenville, North Carolina
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Washington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Akron, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Allentown, Pennsylvania
  - Local Institution, Lancaster, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, West Reading, Pennsylvania
  - Local Institution, York, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Columbia, South Carolina
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Corpus Christi, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, El Paso, Texas
  - Local Institution, Fort Worth, Texas
  - Local Institution, Harlingen, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Tyler, Texas
  - local Institution, Fairfax, Virginia
  - Local Institution, Newport News, Virginia
  - Local Institution, Norfolk, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Roanoke, Virginia
  - Local Institution, Olympia, Washington
  - Local Institution, Seattle, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, La Crosse, Wisconsin
  - Local Institution, Madison, Wisconsin
  - Local Institution, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Local Institution, Ponce
  - Local Institution, Rio Piedras